CLINICAL TRIAL: NCT05589649
Title: Ultrasound-guided Erector Spinae Plane Block Versus Ultrasound-guided Thoracic Paravertebral Block in Pediatric Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Erector Spinae Versus Paravertebral in Pediatric PCNL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP versus Paravertebral
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Renal Stone; Percutaneous; Nephrolithotomy
Keywords: paravertebral block; Erector spinae plane block; Percutaneous nephrolithotomy; pediatric
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental): Ultrasound-guided erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- Paravertebral (Experimental): Ultrasound-guided thoracic paravertebral block
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound-guided erector spinae plane block
  Arms: Erector spinae plane block
Procedure: Paravertebral block — Ultrasound-guided paravertebral block
  Arms: Paravertebral

SUMMARY:
To compare the efficacy of ultrasound-guided erector spinae plane block versus ultrasound-guided paravertebral block in pediatric patients undergoing percutaneous nephrolithotomy

DETAILED DESCRIPTION:
Percutaneous Nephrolithotomy (PCNL) is a commonly performed surgical procedure for complex upper renal tract calculi. Although the skin incision for PCNL appears small, the intensity of intraoperative and postoperative pain is significant owing to soft tissue injury.

Erector spinae plane (ESP) block is an interfascial block that was first described by Forero et al. in 2016. It can be performed by injecting the local anesthetic in the deep interfascial plane of the erector spinae muscle to provide both visceral and somatic analgesia with a sensory level from T2-4 to L1-2.

. Paravertebral block is the technique of injecting local anesthetics in a space immediately lateral to where the spinal nerves emerge from the intervertebral foramina. This technique is used increasingly for intra-operative and post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous nephrolithotomy

Exclusion Criteria:

* Coagulation disorders
* Infection at the site of injection
* Allergy to the local anesthetics used
* Spinal cord abnormalities or neurological deficits

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Total consumption of nalbuphine | The first 24 hours postoperatively
Time to first rescue analgesia | The first 24 hours postoperatively

SECONDARY OUTCOMES:
The concentration of sevoflurane in percent | Through the surgery, an average of 2 hours
Systolic, diastolic, and mean blood pressure during surgery in mmHg | Through the surgery, an average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt